CLINICAL TRIAL: NCT07012187
Title: The Effect of Using Virtual Reality in Subcutaneous Injection Education on the Knowledge and Skills of Nursing Students: A Randomized Controlled Trial
Brief Title: The Effect of Using Virtual Reality in Subcutaneous Injection Education on the Knowledge and Skills of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, BETUL SAHIN KILINC, Lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17162298600-229
Record Dates: First submitted 2025-05-06; First posted 2025-06-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Nursing Education; Nursing Education Research; Virtual Goggles; Virtual Reality
Keywords: nursing education; virtual reality; virtual goggles; nursing skill

STUDY DESIGN:
Intervention Model Description: This study includes experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality- Intervention Group (Experimental): Students will watch a video on subcutaneous injection application using virtual reality technology (virtual reality glasses).
  Interventions: Other: They will watch a video on subcutaneous injection application using virtual reality technology (virtual reality glasses).
- Traditional teaching method-control group (No Intervention): Students will be trained to perform subcutaneous injections using the traditional teaching method.

INTERVENTIONS:
Other: They will watch a video on subcutaneous injection application using virtual reality technology (virtual reality glasses). — Students will watch a video on subcutaneous injection application using virtual reality technology (virtual reality glasses).
  Arms: Virtual Reality- Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate whether virtual reality (VR)-based education improves nursing students' knowledge and skill levels related to subcutaneous injection. The study will include first-year nursing students. The main questions it aims to answer are:

Does the use of virtual reality technology increase knowledge about subcutaneous injection compared to traditional education?

Does virtual reality training enhance practical skill performance in subcutaneous injection?

Researchers will compare a VR-based education group (Intervention Group) with a traditional education group (Control Group) to see if VR education leads to greater improvements in knowledge and skill acquisition.

Participants will:

Complete a knowledge test, a skill test, and a demographic data form before and after the training.

In the Intervention Group, watch a video on subcutaneous injection using VR glasses.

In the Control Group, receive standard education using traditional teaching methods.

Undergo knowledge and skill assessment following the educational interventions.

ELIGIBILITY:
Inclusion Criteria:

* Being a first year student in a nursing undergraduate program.
* Having a health condition and cognitive capacity suitable for using virtual reality technology.
* Having accepted to participate in the study voluntarily.

Exclusion Criteria:

* To give up participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Knowledge level about subcutaneous injection | Before watching videos with virtual reality glasses and 3 weeks after watching videos with virtual reality glasses.
  An information form containing 20 multiple choice questions will be used to measure the level of knowledge about subcutaneous injection. A maximum of 100 points can be obtained from this test forum.
skill performance level about subcutaneous injection | Before watching videos with virtual reality glasses and 3 weeks after watching videos with virtual reality glasses.
  A skill checklist will be used to measure the skill level in subcutaneous injection application. This checklist consists of 25 steps.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I attach importance to the confidentiality of personal data.

REFERENCES:
- [Result] Choi J, Thompson CE, Choi J, Waddill CB, Choi S. Effectiveness of Immersive Virtual Reality in Nursing Education: Systematic Review. Nurse Educ. 2022 May-Jun 01;47(3):E57-E61. doi: 10.1097/NNE.0000000000001117. Epub 2021 Oct 12. PMID 34657101